CLINICAL TRIAL: NCT03969602
Title: The Impact of Cognitive Behavioral Therapy (CBT) on Treatment Outcome After Lumbar Spinal Fusion Surgery in Patients With High Pain Catastrophizing: a Two-center Randomized Controlled Trial of CBT vs. Education Plus Usual Care
Brief Title: Cognitive Behavioral Therapy (CBT) After Lumbar Spinal Fusion in Patients With High Pain Catastrophizing
Acronym: TRIBECA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurocenter of Southern Switzerland (Other)
Collaborators: Maastricht University (Other); Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Pietro Scarone, Staff Neurosurgeon, Principal Investigator, Neurocenter of Southern Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSI-TD/NCH-01
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Spondylolisthesis; Lumbar Instability; Spinal Disease
Keywords: Pain Catastrophizing; Cognitive Behavioral Therapy; Rehabilitation; Spinal disease; Spinal fusion
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Spinal Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigators and research assistants assessing outcomes will be blinded to group assignment. The psychologist/s delivering the CBT and the clinicians delivering the educational intervention in the control group cannot be blinded. Nevertheless, patients will be blinded to study hypotheses and will be informed that the study is examining the comparative benefits of two treatments that are given in addition to usual care and that may potentially improve outcomes. The patients will not be aware of the study hypotheses and will not be informed about the likely association between a high PCS score and lower outcomes after lumbar spinal surgery, neither about the fact that the control intervention (i.e. an educational & exercise intervention that is expected to minimize/cancel any expectation bias) will not address catastrophizing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Participants randomized will receive six individual 1-hour sessions of CBT: two sessions before the operation and four after, delivered by a psychologist trained in CBT for chronic pain. The CBT intervention is tailored to reduce pain catastrophizing. Main techniques are: pain education and the influence of cognitions, emotions and behavior on pain and pain disability; identification of catastrophizing cognitions and replacing them with more adaptive cognitions; stress/anxiety reduction by diaphragmatic breathing and progressive muscle relaxation; emotion regulation skills training; cognitive restructuring; coping skills training to combat helplessness and foster a sense of control and self-efficacy for dealing with acute post-operative pain. The four postoperative sessions build on and further extend the skills learned preoperatively. Each session ends with specific homework assignments. All patients receive a homework book and an individually tailored instruction manual.
  Interventions: Behavioral: Cognitive-behavioral Therapy
- Control Group (Active Comparator): Participants will have six meetings with members of the research team (in person or through telephone). In a first preoperative meeting a member of the team provides verbal information on the preparation for surgery, surgery itself and recovery from surgery, stressing the importance of postoperative exercise. Any questions raised by the patient are discussed. A booklet is provided with information about: structure of the spinal column and spinal diseases; examinations before surgery; the operative environment; surgical procedures; anesthetic procedures; postoperative care and postoperative pain reduction. A second preoperative (telephone) meeting is scheduled to answer any remaining questions. During the postoperative phase, instructions and an exercise manual are provided, Patients keep a diary to record their training activity. Three, six and eight months after discharge patients are contacted by telephone and their training progress is discussed.
  Interventions: Other: Biomedical and surgery-specific education
- Observational Group (low catastrophizing) (No Intervention): Patients will be routinely prescribed medications for pain control and are referred for physical therapy on an out-patient basis in different sites or an in-patient basis in specialized rehabilitation centers following lumbar spinal fusion surgery, depending on the needs. Typically, a full rehabilitation regime starts 2-3 weeks after surgery. Usual programs involve active spinal mobilization aimed at gradually improving the range of motion, exercises to strengthen spinal deep muscles, and segmentary stretching involving the lower limb and back muscles, together with manual therapy. The patients are also given walking exercises and trained in how to change position.

INTERVENTIONS:
Behavioral: Cognitive-behavioral Therapy — The biopsychosocial approach of CBT focuses on the complex interaction between psychological, social and biological factors. The biopsychosocial model assumes that health problems are hardly ever limited to just one domain of human experience but by multiple domains of human experience. CBT helps patients understand thoughts and feelings that influence behaviors. It consists of a cognitive aspect and a behavioral aspect. The cognitive aspect is based on Becks cognitive model: the way that individuals perceive a situation is more closely connected to their reaction than the situation itself. A person's cognition has impact on their mood and emotions, their bodily reactions and their behavior. The second part of cognitive behavior therapy focuses on the actual behaviors that are contributing to the problem. The goal of CBT is to identify maladaptive thoughts and change them into more realistic and constructive thoughts to modify feelings and behavior and thereby the experience of pain.
  Other Names: CBT
  Arms: Experimental Group
Other: Biomedical and surgery-specific education — Biomedical and surgery-specific education preoperatively and an exercise manual postoperatively.
  Arms: Control Group

SUMMARY:
Catastrophizing has emerged as the strongest independent predictor for persistent postsurgical pain. Although behavioral interventions, including Cognitive Behavioral Therapy (CBT), have been shown to reduce the impact of persistent pain, postsurgical patients have not historically been offered these interventions. The aim of our study is to examine whether an intervention targeting pain catastrophizing can reduce the risk of persistent pain and disability after spinal fusion.

Our primary hypothesis is that a perioperative cognitive behavioral intervention with the goal to decrease anxiety and pain catastrophizing will decrease the risk of persistent pain and disability after spinal fusion surgery in high catastrophizing patients.

To study this hypothesis the investigators will perform a prospective, randomized, controlled multicenter trial with 1:1 allocation, comparing 2 cohorts.

Patients aged > 18 years/old, with a primary diagnosis of spinal stenosis, degenerative or isthmic spondylolisthesis or degenerative disc disease (DDD) determined by expert spine surgeons and selected for lumbar spinal fusion surgery with decompression will be screened for high levels of pain catastrophizing using the Pain Catastrophizing Scale (PCS). Patients with a score of ≥ 24 on the PCS who will consent to the study will be randomized to CBT (2 sessions preoperatively and 4 sessions postoperatively) plus usual care (experimental group) or usual care (control group). To limit expectation bias, an educational intervention will be added in the control group.

Primary outcome is the Core Outcome Measure Index (COMI) at 12 months. Secondary outcomes are scores on 11-point Numeric Rating Scale (NRS) for back and leg pain, Oswestry Disability Index (ODI), Patient-reported outcomes measurement - depression (PROMIS-D), Patient Global Impression of Change (PGIC), Pain Catastrophizing (PCS), reliance on analgesics and employment status. NRS will be measured on the 4th postoperative day, at 8 weeks, 6 months and 1 year, while all other outcomes will be measured at 8 weeks, 6 months and 1 year.

DETAILED DESCRIPTION:
The incidence of moderate to severe chronic postsurgical pain (CPSP) at 12 months after surgery is circa 12% in Europe, depending in part upon the surgical procedure. Worldwide, more than 230 million people undergo major surgery every year; the global annual cost of new cases of CPSP is in the hundreds of billions of dollars. The response to this costly tragedy has been unacceptably slow.

Perioperative protocols have historically not incorporated routine screening for patients at-risk for post-surgery persistent pain or compromised function. However, early detection and management of patients at high risk for CPSP may modify the postsurgical pain trajectory and reduce the incidence of CPSP.

In particular, persistent pain and disability after spinal surgery poses a large problem. Around 20% of the patients have persistent or recurrent pain in the back or limbs after surgical interventions for spinal disease. Several risk factors for such unfavorable outcomes have been identified, among which psychological factors. The most robust psychological predictors of high levels of acute postsurgical pain and of persistent pain in the back or limbs after spinal surgery are high levels of preoperative anxiety and pain catastrophizing.

Psychological variables are modifiable and could be target for intervention. Cognitive Behavioral Therapy (CBT) is the leading psychological treatment for chronic pain. CBT aims to reduce maladaptive cognitions and behaviors and replace these with more adaptive ones. CBT has been shown to reduce anxiety and catastrophizing and to increase self-efficacy and feelings of control beliefs and through this lowers pain-related disability and pain interference (including sleep problems and depression).

This study is a prospective, randomized, controlled multicenter trial with 1:1 allocation, comparing lumbar spinal fusion surgery outcome between 2 groups with high pain catastrophizing, 1 that receives perioperative CBT plus usual care (experimental group) and 1 that receives usual care (control group). To minimize expectation bias in patients, an educational intervention is added in the control group.

Patients will be enrolled in the Department of Neurosurgery at the Neurocenter of Southern Switzerland, Lugano Regional Hospital and the department of Neurosurgery of Zuyderland Medical Center, Heerlen, The Netherlands.

Patients with as score of ≥ 24 on the PCS will be eligible to be randomized to perioperative CBT plus usual care or education plus usual care.

Data collection sessions will occur for each patient randomized, at baseline, at 8 weeks, and at 6 and 12 months following surgery. A third, non-randomized group is also included, consisting of low catastrophizing patients. These patients will not undergo any additional intervention besides usual care, but will undergo the same data-collection as the high catastrophizing randomized groups. This offers the possibility to examine whether CBT can reduce the negative effects of catastrophizing on outcome to the level of improvement one would expect in non-catastrophizing patients. Staff blinded to group assignment will contact patients by phone at circa one week before data collection time points to remind them to fill in the questionnaires.

Primary hypothesis of the investigators is that patients randomized to the CBT group show a greater improvement on the Core Outcome Measures Index (COMI) at 12 months post-surgery compared to patients randomized to the control group.

Secondary hypotheses are that patients randomized to the CBT group show a larger reduction in disability (ODI), leg/back pain (NRS), depression and pain catastrophizing (PCS) at 12 months post-surgery compared to patients randomized to the control group. Moreover, patients in the CBT group report higher global impression of chance, less reliance on analgesics and better employment status compared to patients in the control group. Finally, the investigators hypothesize that the high catastrophizing group receiving the control intervention will have worse outcomes on all measures compared to the low catastrophizing group receiving standard care, whereas the high catastrophizing group receiving the CBT intervention will have comparable outcomes as the low catastrophizing group.

All included patients will be assessed before surgery for the outcomes of interest. Patients assigned to the CBT intervention condition will attend six individual 60-min CBT sessions (2 before and 4 after surgery). Patients randomized to the education condition will receive six session of biomedical education and an exercise program. Non-randomized low catastrophizing patients do not receive an additional intervention. All patients will receive care that they would have routinely received had they not been entered in the study (i.e. standard postoperative physical therapy). The three groups of patients will undergo the same data collection procedures.

The primary outcome is the difference in the COMI between the study groups, 12 months after surgery. A difference of two points is considered clinically meaningful [44]. With an assumed SD of 2.5, the effect size of this difference, quantified as Cohen's d is 0.80. Inclusion of 42 patients per intervention group will yield a power of 0.95 at a type-I error rate of 0.05. In addition, 42 patients with low pain catastrophizing scores will undergo the same assessments, but not receive any intervention besides care as usual. Taking into account a drop-out rate of 15%, 150 patients will be included in total.

Baseline patient characteristics will be stratified by group and presented as mean and standard deviation (SD), median and first and third quartile, and count and percentage, as appropriate. Differences in baseline characteristics between randomized groups will not be statistically tested, whereas differences with the separate control cohort will be tested using the independent-samples t-test for continuous variables, and Pearson's chi-square test for categorical variables. In case of expected cell counts of less than 5, Fisher's Exact test will be used instead.

All patients randomized (i.e. those with a PCS score > 24) will be analyzed in an intention-to-treat analysis. To test for a difference between the CBT and control group in the COMI at 12 months, linear regression will be used, with correction for baseline COMI and center. In addition, the difference in the trajectory of COMI over time will be assessed by means of linear mixed-effects regression, taking all follow-up measurements into account. Adjustment for center, type of surgery, age and gender will be made and, if necessary, for other prognostic variables significantly associated with the outcome (i.e., acute postoperative pain intensity, preoperative depression, preoperative surgical fear, length of current sick leave, pain duration). Stepwise backward elimination using the Wald test will be used to select prognostic variables significantly associated with the outcome. Any control variables that are incomplete will be imputed if the proportion of incomplete patients exceeds 0.05. Investigators will use multiple imputation with fully conditional specification with the number of imputations set to the percentage of incomplete patients. Predictive mean matching will be used to draw values to be imputed. Secondary outcome variables will be analyzed similar to the primary outcome. For these, logistic regression analysis adjusted for center will be used to test for differences in proportions at 12 months postoperatively.

Exploratory, investigators will compare the outcomes of the patients in the two intervention groups with the outcomes of patients with low pain catastrophizing scores (i.e. those with a PCS score < 24) undergoing care as usual. Linear mixed-effects regression for the three groups will be performed with primary and secondary outcomes at the three postoperative assessment periods and controlling for preoperative values. This analysis will indicate whether high catastrophizing patients follow a similar trajectory of pain and functioning after spinal fusion surgery compared non-catastrophizing patients.

ELIGIBILITY:
Inclusion Criteria:

* able to read and speak Italian (site 1) or Dutch (site 2)
* a primary diagnosis of spinal stenosis, degenerative or isthmic spondylolisthesis or degenerative disc disease (DDD) determined by expert spine surgeons
* selected for lumbar spinal fusion surgery with decompression
* patients with a score of ≥ 24 on the PCS to be randomized to perioperative CBT plus usual care or education plus usual care, required to complete all questionnaires (see study schedule)
* patients with a score of < 24 will not be randomized to one of the treatment groups but are eligible for preoperative and postoperative assessment
* are able to provide informed consent and have signed the informed subject consent form

Exclusion Criteria:

* report plans to undergo major surgery within six months after current lumbar spinal fusion surgery
* comorbid severe psychiatric conditions
* known or suspected non-compliance, drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to dementia, etc. of the participant
* the presence of any serious medical comorbidity such as sepsis or cancer that might cause disability or worsen the patient's general health condition
* pregnancy is an "automatic" exclusion because women who are pregnant are excluded by their physicians from lumbar spinal fusion surgery
* an opioid intrathecal pump
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
COMI (Core Outcome Measure Index) | 12 months post surgery
  The COMI comprises a short set of questions used to assess the impact of spinal disorders on multiple patient-orientated outcome domains. It is based on a set of individual items selected from established questionnaires and recommended for standardized use by an international group of experts in the field. It consists of seven items to assess the extent of the patient's back pain and leg pain, difficulties with functioning in everyday life, symptom-specific well-being, general quality of life, and social and work disability. A summary index score from 0 (best health status) to 10 (worst health status) can be computed by averaging the values of the five subscales.

SECONDARY OUTCOMES:
NRS Pain (The Numeric Rating Scale for Pain) | 4 days, 8 weeks, 6 and 12 months post surgery
  NRS-11 is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. Rating = 0 indicates no pain, rating =1-3 indicates mild pain, rating 4-6 indicates moderate pain while rating 7-10 indicates severe pain.
ODI (Oswestry Disability Index) | 8 weeks, 6 and 12 months post surgery
  The ODI questionnaire is a self-administered set of ten questions assessing the patient's level of pain and function during activities of daily living such as walking, personal care, standing, sleeping, etc. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score as follows: 0%-20%=Minimal disability, 20%-40% = Moderate disability, 40%-60% = Severe disability, 60%-80%= Crippled, 80%-100% = bed bound.
PROMIS (Patient-Reported Outcomes Measurement Information System) for depression | 8 weeks, 6 and 12 months post surgery
  The PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. For the present study, the PROMIS Short Form v1.0 - Depression 8b will be used. This questionnaire, part of the PROMIS depression toolbox, has 8 items that are scored on a 1- 5 scale. For each question, a score of 1 indicates "never" (better score) while a score of 5 indicates "always" (worse score). A total score is obtained by summing the values of the responses to each question, ranging from 8 (low level of depression) to 40 (high level of depression).
PGIC (Patient's global impression of change) | 8 weeks, 6 and 12 months post surgery
  Patients rate their perceived improvement on a 7-point Likert Scale from 1 (very much improved) to 7 (very much worse).
PCS (Pain catastrophizing) | 8 weeks, 6 and 12 months post surgery
  The Pain Catastrophizing Scale (PCS) has 13 items that are scored on a 5-point scale ranging from 0 (never) to 4 (always), providing a total score that can range from 0 to 52.
EQ-5D-5L (The 5-level EuroQol 5 Dimensions) for quality of life | 8 weeks, 6 and 12 months post surgery
  The EQ-5D-5L questionnaire uses a health state classification defining health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems and 5= extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state, ranging from 11111 (no problems in any of the 5 dimensions) to 55555 (extreme problems in all dimensions). The health states are then converted into a single index value from 0 (worse) to 1 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Scarone, M.D., Principal Investigator — Neurocenter of Southern Switzerland
Locations (1):
- Neurocenter of Southern Switzerland, Neurosurgical Service, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scarone P, Smeets AYJM, van Kuijk SMJ, van Santbrink H, Peters M, Koetsier E. A randomized controlled TRIal of cognitive BEhavioral therapy for high Catastrophizing in patients undergoing lumbar fusion surgery: the TRIBECA study. BMC Musculoskelet Disord. 2020 Dec 4;21(1):810. doi: 10.1186/s12891-020-03826-w. PMID 33276768